CLINICAL TRIAL: NCT04257760
Title: Understanding Palliative Care and End of Life Needs in the ALS Population: The First Step to Improving Patient and Caregiver Quality of Life
Brief Title: Evaluation of Palliative Care for Patients With ALS and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: ALS Society of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALSPall1
Record Dates: First submitted 2020-01-17; First posted 2020-02-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; palliative care; caregivers
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: It is a pilot trial to assess the feasibility of palliative care for ALS patients. Patients will be in the palliative care or non-palliative care arm of the trial based on their decision to have a palliative care consultation or not. If they do not initially chose a palliative care consult they can change their mind during the course of the trial.
Masking Description: The patients, the palliative care physicians and the research team will know if a palliative care consultation has been done or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): These ALS patients and their caregivers will receive standard care.
- Early palliative care (Experimental): These patients will receive a palliative care consultation that would not be requested by their care team as standard of care.
  Interventions: Behavioral: Palliative Care consultation outside standard of care

INTERVENTIONS:
Behavioral: Palliative Care consultation outside standard of care — The ALS patients and their caregivers will receive a consultation with a palliative care physician. This will take approximately one hour and occur in their location of choice (ie. often the patient's home). Subsequent palliative care consultations will occur at the discretion of the ALS patient and the palliative care physician.
  Arms: Early palliative care

SUMMARY:
Rationale: Amyotrophic lateral sclerosis (ALS) is a degenerative illness which currently has no medical cure. It is routinely accompanied by a significant symptom burden including high levels of distress in patients and their caregivers. As a result, an early palliative care approach is recommended in the ALS population. Palliative care has been shown to have positive effects on the quality of life in patients and caregivers in other life limiting illness such as cancer and multiple sclerosis. Unfortunately, our understanding of the palliative care needs in ALS is limited and the efficacy of palliative care involvement is poorly understood. Furthermore, ALS patients are largely underserved by palliative care in Ontario, with <50% of ALS patients receiving palliative care even in the last year of life. Hypothesis: The investigators hypothesize that ALS patients will be agreeable to palliative care consultations and that this will improve the quality of life of patients and their caregivers. Specific Aims: This project seeks to initiate routine palliative care consultation in an interdisciplinary ALS clinic to: 1) improve patient and caregiver quality of life, 2) further understand the palliative care needs of the ALS population and 3) identify which patients and caregivers are most likely to benefit from palliative care consultation, thus guiding clinicians on when to refer in the future. Significance: This study is the first investigate the feasibility and efficacy of palliative care consultation in the ALS population, and its effects on quality of life. It has the potential to provide increased support to patients as well as caregivers. Finally, this study will aid in our understanding of the optimal time to involve palliative care in the ALS population and will act as a foundation on which larger, controlled studies can be built.

DETAILED DESCRIPTION:
Patient recruitment:

Patients who are eligible for the study will be asked by their ALS care team if they would like to speak to the research assistant about the study. Patients may also self refer if they hear about the study and are interested in learning more about it. As a part of this study, participants will meet briefly with a palliative care (PC) physician to discuss the goals of palliative care and the interventions a palliative care physician can provide. As part of the study, patients will be offered the choice of a palliative care consultation (in a timely manner - either at home or at the ALS clinic) or no palliative care consultation. Participants will fill out a brief questionnaire regarding their interest in a PC consultation. Relevant demographic information such as time since diagnosis and functional ability will be collected for all patients included in the study. This study is planned to recruit patients for the period of one year, with a total study period of 18 months (i.e. the first patient included to the study will be followed until death or for 18 months and the last patient recruited to the study will be followed for 6 months).

Outcome Measures:

All patients who agree to participate in the study, will be asked to complete two scales which measure quality of life: The ALS Specific Quality of Life Revised Scale (ALSSQOL-R,) a validated instrument to measure quality of life in ALS patients (8, 15) and the Hospital Anxiety and Depression Scale (HADS), a validated instrument for measuring anxiety and depression in patients and caregivers(16). These scales will be completed at baseline, 1 month, 3 months and every 3 months for the entirety of the study period. Caregivers will complete the HADS at the same time interval. The ALSSQOL-R and HADS require 10-20 minutes and 2-5 minutes to complete, respectively (15, 17). The ALSSQOL-R is routinely used as pre-visit screening in multidisciplinary ALS clinics and is felt to be feasible in the ALS population(15). The invitation to the study and coordination of survey completion will be led by a research assistant and not a member of the patient's care team. Survey completion rates and feasibility of routine completion will be examined. Qualitative reasons for declining a PC consult at the time of study initiation, as reported by patients on the consent to PC consultation questionnaire, will also be recorded.

Patients and caregivers who receive a PC consult as a part of the study period will complete a questionnaire focusing on their satisfaction with the consultation, its timeliness (i.e. too early or too late in their illness trajectory) and any fatigue or distress which resulted from the consultation. Follow-up PC assessments will occur as determined by the patient and PC physician. Patients and caregivers who decline participation in the study as well as those who are included in the study but declined PC consultation will continue with usual care and thus be referred to a PC specialist at the discretion of their physicians. A detailed overview of the plan for study recruitment and planned outcome measures are outlined in Figure 1 and Table 1.

Analyses Strategy:

This study will focus on several different outcomes as listed in Table 1. The main outcome will be the effect of PC consultation on patient and caregiver quality of life. This will be determined by evaluating a change in ALSSQOL-R and HADS scores in patients and caregivers over time, both individually and between the groups of patients who received and did not receive a PC consult. Unfortunately, there are no previously reported minimally important differences for these scales in the ALS population. Difference in quality of life indicators will be examined between patients who received PC involvement and those in the usual care group. Mean quality of life scores will be compared at different time points post consultation and statistical significance will be determined using t-tests. Quality of life scores pre and post palliative care consultation will also be examined in patients and caregivers at different time points. They will be reported as mean scores (+95% confidence intervals) and significant change will be determined using univariate analyses. As this study has a focus on describing the PC needs of the ALS population, chart reviews of PC consults will be completed to identify the major themes and issues discussed in PC consults.

Process measures for this study will also be examined. These include the proportion of patients that were approached who consented to be in the study, proportion of patients in the study who choose a PC consultation, the duration of the PC consultation, the number of follow-up appointments per patient, the delay between enrollment in the study and initial PC consultation. The acceptability and satisfaction with PC involvement will be assessed by qualitative and quantitative measures including patient and caregiver self-reported reasons for accepting or declining a PC consultation and responses to post PC satisfaction questionnaire. Balancing measures and potential negative effects of PC consultation, including anxiety and fatigue, will be assessed via the post PC consultation satisfaction scale. If data allows, subsequent studies may focus on the change in health care utilization (i.e. emergency department visits, hospitalizations etc.) in the group of patients who received PC when compared to the usual care group.

Given the variability in presentation and often rapid clinical decline experienced by patients with ALS, the idea of early PC for all patients is likely not feasible and unlikely to be beneficial. Some patients may experience significant impairment and the time of diagnosis and benefit from immediate referral, while others may experience a period of stability and be comfortable without referral. Considering this, a goal of this study is understanding which factors are most likely to prompt a referral to PC, and which patients are most likely to benefit from a PC referral. As a part of the study, PC consultations and patient records will be reviewed and demographic information such as ALS Functional Rating Scale score (ALSFRS -R), time since diagnosis and the presence or absence of symptoms will be considered. This will be linked to reported quality of life scores to identify which factors are most likely to improve with PC referral and which factors are most associated the need for PC referral. This will help guide clinicians nationwide as to when to consider PC referrals in their patients, with the goal of ensuring patients have timely access to PC at the appropriate time.

Potential Impact:

Ultimately, there is immense potential to improve patient quality of life with this project. It is the first to introduce routine PC into a multi-disciplinary ALS clinic in Ontario, a population that is largely underserviced by PC. It seeks to understand the physical and emotional factors which limit patient quality of life and links to physicians and resources to act on these issues. This project also plans to improve the quality of life of caregivers, providing increased support and further understanding of caregiver needs. The investigators hope to identify the factors that make a patient/caregiver most likely to benefit from PC; which will guide referral criteria for all patients with ALS and ensure that PC consultations are available to patients at a timely manner when it is most likely to be impactful. Finally, this study will improve the capacity of current health care providers to address patient and caregiver quality of life concerns. It will provide a new foundation of knowledge on which larger, controlled studies can be built in the future.

ELIGIBILITY:
Inclusion Criteria:

Patient with ALS at the Ottawa Hospital ALS clinic or caregiver of participating patient.

Exclusion Criteria:

Significant cognitive impairment Prior palliative care consultation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in average ALS Specific Quality of Life - Revised score in ALS patients post palliative care | At baseline compared to 1 month and 3 months after palliative care consultation
  the change in the average score of ALS patients on the ALS Specific Quality of Life - Revised scale. On the scale the minimum score is 0 and the maximum score is 460. A higher score reflects a higher quality of life.
Difference in average ALS Specific Quality of Life - Revised score between arms | At baseline, 1 month and 3 months after palliative care consultation or study enrollment
  The difference between the average ALS Specific Quality of Life - Revised score between ALS patients who received the palliative care consultation and patients who did not. On the ALS Specific Quality of Life - Revised scale the minimum score is 0 and the maximum score is 460. A higher score reflects a higher quality of life.
Difference in average Hospital Anxiety and Depression Scale score for ALS patients between arms | At baseline, 1 month and 3 months after palliative care consultation or study enrollment
  The difference between the average Hospital Anxiety and Depression Scale score between ALS patients who received the palliative care consultation and patients who did not. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.
Difference in average Hospital Anxiety and Depression Scale score for caregivers of ALS patients between arms | At baseline, 1 month and 3 months after palliative care consultation or study enrollment
  The difference between the average Hospital Anxiety and Depression Scale score between caregivers of ALS patients who received the palliative care consultation and caregivers of patients who did not. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.
Change in average Hospital Anxiety and Depression Scale score in patients with ALS | At baseline compared to 1 month and 3 months post palliative care consultation
  the change in the average Hospital Anxiety and Depression Scale scores in ALS patients. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.
Change in average Hospital Anxiety and Depression Scale score in caregivers of patients with ALS | At baseline compared to 1 month and 3 months post palliative care consultation
  The change in the average Hospital Anxiety and Depression Scale scores for caregivers of ALS patients. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.

SECONDARY OUTCOMES:
Patient satisfaction with palliative care consultation on the Satisfaction with Palliative Care Questionnaire | at 24 months
  description of the average scores for questions on the Palliative care satisfaction.questionnaire. The minimum score is 9 and the maximum score is 45. A higher score indicates greater satisfaction with palliative care.
care provided through palliative care consultation | at 24 months
  description of type and frequency of issues covered as part of the palliative care consultation and the palliative care interventions provided
reasons for decision to pursue palliative care consultation or not | at 24 months
  description of the reasons patients list for pursuing or not pursuing palliative care consultation as well as the frequency of each reason
Change in average ALS Specific Quality of Life - Revised score in ALS patients post palliative care | At baseline compared to 6 month, 12 months, 15 months, 18 months, 21 months after palliative care consult
  the change in the average score of ALS patients on the ALS Specific Quality of Life - Revised scale. On the ALS Specific Quality of Life - Revised scale the minimum score is 0 and the maximum score is 460. A higher score reflects a higher quality of life.
Change in average Hospital Anxiety and Depression Scale score in ALS patients post palliative care | At baseline compared to 6 month, 12 months, 15 months, 18 months, 21 months after palliative care consult
  the change in the average score of ALS patients on the Hospital Anxiety and Depression Scale. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.
Change in average Hospital Anxiety and Depression Scale score in caregivers of ALS patients post palliative care | At baseline compared to 6 month, 12 months, 15 months, 18 months, 21 months after palliative care consult
  the change in the average score of caregivers of ALS patients on the Hospital Anxiety and Depression Scale. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.
Difference in average ALS Specific Quality of Life - Revised score between arms | at 6 months, 12 months, 15 months, 18 months, 21 months after palliative care consultation or study enrollment
  The difference between the average ALS Specific Quality of Life - Revised score between ALS patients who received the palliative care consultation and patients who did not.On the ALS Specific Quality of Life - Revised scale the minimum score is 0 and the maximum score is 460. A higher score reflects a higher quality of life.
Difference in average Hospital Anxiety and Depression Scale score between arms in ALS patients | at 6 months, 12 months, 15 months, 18 months, 21 months after palliative care consultation or study enrollment
  The difference between the average Hospital Anxiety and Depression Scale score between ALS patients who received the palliative care consultation and patients who did not.The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.
Difference in average Hospital Anxiety and Depression Scale score between arms in caregivers of patients with ALS | at 6 months, 12 months, 15 months, 18 months, 21 months after palliative care consultation or study enrollment
  The difference between the average Hospital Anxiety and Depression Scale score between caregivers of ALS patients who received the palliative care consultation and patients who did not. The minimum for depression or anxiety is 0. The maximum score for depression or anxiety is 21. The higher the score, the more pronounced the symptoms.

OTHER OUTCOMES:
Proportion of patients who complete a palliative care consultation | at 24 months
  The number of patients who choose to have a palliative care consultation as part of the study divided by the total number of patient participants

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn C Zwicker, MD, Principal Investigator — The Ottawa Hospital; Christine Watt, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watt CL, Smith IC, Rice J, Murphy R, Breiner A, Duff MLV, Nogo D, Bush SH, McNeely S, Buenger U, Zehrt B, Zwicker J. Qualitative Analysis of Initial Palliative Care Consultations in Amyotrophic Lateral Sclerosis. J Pain Symptom Manage. 2024 Jul;68(1):43-52.e2. doi: 10.1016/j.jpainsymman.2024.03.024. Epub 2024 Apr 2. PMID 38574876
- [Derived] Zwicker J, Smith IC, Rice J, Murphy R, Breiner A, McNeely S, Duff M, Buenger U, Zehrt B, Nogo D, Watt CL. Palliative care at any stage of amyotrophic lateral sclerosis: a prospective feasibility study. Front Med (Lausanne). 2023 Sep 13;10:1204816. doi: 10.3389/fmed.2023.1204816. eCollection 2023. PMID 37780560